CLINICAL TRIAL: NCT07259174
Title: Ultrasound of the Diaphragm Excursion Ratio as Physiological Biomarker in Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Acronym: Undated 2
Status: Recruiting | Type: Observational
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Wytze de Boer, MD, University Medical Center Groningen
Other Study IDs: Diaphragm 003
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: COPD
Keywords: diaphragm; ultrasound; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Study group will receive ultrasound of the diaphragm on admission for acute exacerbation COPD. No further study interventions.

SUMMARY:
3.1 Introduction and rationale In 2020 an estimate of 562.700 people had Chronic Obstructive Pulmonary Disease (COPD) in the Netherlands, resulting in 21.335 hospital admissions.[1] An acute exacerbation COPD (AECOPD) in combination with hospital admission is associated with high mortality and morbidity. [2]

Noninvasive ventilation (NIV) has been very effective in the context of AECOPD, since it efficiently offloads respiratory muscles and counteracts dynamic hyperinflation. This method often prevents intubation as a bridge to administering effective therapies (e.g., glucocorticoids, bronchodilators, and antibiotic agents)[3], and may reduce mortality.[4] Current guidelines recommend NIV for the treatment of acute respiratory failure in patients with respiratory distress, pH < 7.35, and PaCO2 > 6 kPA (with exclusion of patients requiring invasive ventilation, see guideline).[5,6] National guidelines do not recommend NIV in AECOPD with increased work of breathing without respiratory acidosis due to lack of evidence. [5]

Ultrasound of the diaphragm can identify atrophy and impaired motion or contractility of the diaphragm[10], and has been shown to predict mortality and NIV failure during NIV treatment for respiratory acidosis due to AECOPD.[11-15] Whether ultrasound of the diaphragm may predict mortality or need for (non-)invasive ventilation in AECOPD without respiratory acidosis on initial presentation is unknown.

During exploratory analysis of a previous study (unpublished; NCT05671198) we might have found a marker that has the potential to predict progression to NIV or death during hospitalization for AECOPD without respiratory acidosis:

The difference between diaphragm motion during tidal breathing and maximal breathing, used as a surrogate for inspiratory reserve volume (IRV), was significantly lower in patients requiring NIV or who died in-hospital compared to those who did not (1.59 cm, SD 1.91 vs. 3.14 cm, SD 2.45; p = 0.033). We performed a ROC curve analysis to assess the predictive value of these variables, which yielded an area under the ROC curve (AUROC) of 0.752 (95% CI: 0.535 - 0.968, p = 0.033), indicating a statistically significant discriminatory ability. The best cut-off value, as determined with the Youden's J statistic, was 1.74 cm, with a sensitivity of 86% and specificity of 70% for predicting NIV requirement or inhospital death.

However, the number of events was low and the study was primarily powered for another outcome. Therefore, prospective validation is needed before we impose treatment based on this marker. In case the suggested ultrasound measurement (see introduction) proofs to be a discriminatory marker for deterioration during hospitalization or predictive of progression to Non-Invasive Ventilation, we hope to be able to perform a follow-up study in which patient will be randomized to either standard of care or 'elective' NIV (to avoid emergency NIV need) based on yet to determine cut-off values.

3.2 Design (including population, method, confounders and outcomes) A multi-center, prospective observational cohort study conducted at Isala Hospital and UMCG aimed at determining the value of the sonographic motion ratio (tidal/maximum) of the diaphragm in AECOPD after hospital admission. After enrollment, the sonographic diaphragm motion will be assessed as additional measurement during standard-of-care lung ultrasound (POCUS), after which hospital outcomes will be registered. Primary outcome will be the sensitivity of this ultrasound marker for in-hospital deterioration (progression to NIV of death). Secondary analysis will include predictive models.

3.3 Research question What is the sensitivity of the diaphragm motion ratio (tidal/maximum) during ultrasound for in-hospital deterioration (progression to NIV or death) in AECOPD.

DETAILED DESCRIPTION:
See summary

ELIGIBILITY:
• Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Hospitalization primarily because of severe acute exacerbation of COPD
* Spirometry record within last 5 years, with: post-bronchodilator FEV1/FVC < 0,70 and FEV1% < 80%predicted
* Minimum of 10 packyears

  * Exclusion criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Established diagnosis of diaphragm diaphragm paralysis.
* Inability for diaphragm imaging (e.g. mechanical ventilation, or unable to follow vocal instructions).
* Those not able or unwilling to give written informed consent.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized AECOPD patients
Sampling Method: Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
primary outcome | From enrollment to the end of hospitalization
  The primary endpoint is the sensitivity of the diaphragm motion ratio (ultrasound marker) for predicting in-hospital deterioration (defined as progression to non-invasive ventilation or in-hospital death). Sensitivity will be calculated as: True Positives/(True Positives+False Negatives)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Isala, Zwolle, Overijssel
  - University Medical Centre Groningen, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT07259174/Prot_SAP_000.pdf